CLINICAL TRIAL: NCT07181265
Title: A Single-center, Non-randomized, Open-label, Self-controlled Phase I Drug-drug Interaction Clinical Study to Evaluate the Pharmacokinetics of JMKX003142 With Amiodarone, and Febuxostat in Chinese Healthy Subjects
Brief Title: Drug-Drug Interaction of JMKX003142 With Amiodarone and Febuxostat in Healthy Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jemincare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: JMKX003142-103
Record Dates: First submitted 2025-09-12; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease (ADPKD)
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant | interventions — Amiodarone; Febuxostat

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug-Drug interaction study of JMKX003142 and Amiodarone (Experimental): 24 Subjects first administered with JMKX003142 tablets 4mg from day 1 to day 7 after breakfast. from day 12 to day 18 the subjects were adminstered with Amiodarone Hydrochloride Tablets 400 mg. from day 22 to day 28 these subjects were co-adminstered with JMKX003142 tablets 4mg and Amiodarone Hydrochloride Tablets 400 mg.
  Interventions: Drug: Amiodarone Hydrochloride Tablets
- Drug-Drug interaction study of JMKX003142 with Febuxostat (Experimental): 24 Subjects first administered with JMKX003142 tablets 4mg from day 1 to day 7 after breakfast. from day 12 to day 18 the subjects were adminstered with Febuxostat Tablets 40 mg. from day 21 to day 27 these subjects were co-adminstered with JMKX003142 tablets 4mg and Febuxostat Tablets 40 mg.
  Interventions: Drug: Febuxostat Tablets

INTERVENTIONS:
Drug: Amiodarone Hydrochloride Tablets — Cohort 1: The intervention is for study of drug drug interaction of JMKX003142 when administered with Amiodarone
  Arms: Drug-Drug interaction study of JMKX003142 and Amiodarone
Drug: Febuxostat Tablets — Cohort 2: The intervention is for study of drug drug interaction of JMKX003142 when administered with Febuxostat Tablets
  Arms: Drug-Drug interaction study of JMKX003142 with Febuxostat

SUMMARY:
This is a open-label, non-randomized, multiple oral dosings, three-period, drug-drug interaction study of JMKX003142 tablet, Amiodarone Hydrochloride Tablets and Febuxostat Tablets in Chinese healthy adult subjects

ELIGIBILITY:
Inclusion Criteria:

1. Able to participate and comply with all study procedures and restrictions, and willing to provide written informed consent to participate in the study.
2. Healthy adult males and/or females, 18 to 45 years of age (inclusive) at the date of signed consent form. Body mass index (BMI) greater than or equal to 18 and less than 32 (kg/m2) and a minimum body weight of 45 kg.
3. The health of the subjects was determined by the investigator based on medical history, physical examination, clinical laboratory examination, and 12-lead electrocardiogram, all of which were determined by the investigator to be normal or not clinically significant.
4. Women of child-bearing potential and sexually active males willing to use highly effective methods of contraception from screening until 3 months after last dose of study drug. In addition, participants must not donate sperm/egg for the time period specified above.

Exclusion Criteria:

1. Subjects having hypersensitivity to study drug or have a history of allergies to multiple drugs, foods, or other substances
2. History or presence of significant circulatory system, respiratory system, digestive system, blood system, urinary and reproductive system, endocrine and metabolic system, nervous system, mental system, muscular and skeletal system, skin system, lymphatic system, immune system, Otolaryngology or other related systems disease or disorder. as well as systemic or local acute or chronic infections.
3. Subjects with dysphagia, gastrointestinal diseases, or any conditions that may affect drug absorption; such as a history of hepatobiliary and pancreatic diseases, gastrointestinal diseases, gastrointestinal surgery (except appendectomy), or a history of chronic pancreatitis, idiopathic acute pancreatitis, or habitual diarrhea.
4. Vital signs during the screening period meet any of the following conditions: systolic blood pressure >140 mmHg or <90 mmHg; diastolic blood pressure >90 mmHg or <50 mmHg (Cohort 1: diastolic blood pressure >90 mmHg or <60 mmHg); pulse >100 beats/min or <50 beats/min (Cohort 1: pulse >100 beats/min or <60 beats/min); ear temperature >37.5°C or <35°C.
5. History of QTc interval prolongation or abnormal ECG results during screening, QTcF ≥ 450 ms for males or ≥ 470 ms for females, or QRS interval > 120 ms.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-10-30 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Cmax，ss | up to 7 days
AUC0-tau | up tp 7 days

SECONDARY OUTCOMES:
Tmax | up to 7 days
AUC0-t | up to 7 days